CLINICAL TRIAL: NCT05061966
Title: Piloting a Web App for Sexual and Gender Minority Youth Mental Health
Brief Title: The Digital Wellbeing Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: HopeLab Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 849509
Record Dates: First submitted 2021-09-14; First posted 2021-09-30 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Mental Health
Keywords: Sexual and Gender Minorities
MeSH Terms: conditions — Psychological Well-Being; Coitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Resource website (Active Comparator): The comparator is a website that includes a list of freely available web-based resources for sexual and gender minority youth.
  Interventions: Behavioral: Control
- immi (Experimental): The intervention is a novel and scalable web application designed to provide sexual and gender minority youth with tools for affirming their identity and coping with minority stress.
  Interventions: Behavioral: immi

INTERVENTIONS:
Behavioral: immi — The intervention has four main content areas: 1) gender identity (the gender guide), 2) sexual orientation (the queerness guide), 3)stress and coping (the stress guide), and 4) internalized stigma (the internalized stigma guide).
  Arms: immi
Behavioral: Control — The control will have access to resources on the website, but will not receive any engagement reminders, matching the conditions present in real world contexts in which web-based resource lists are available.
  Arms: Online Resource website

SUMMARY:
This goal of this randomized control trial is to test whether a web application that provides sexual and gender minority youth ages 13-19 (N=200) with tools for affirming their identities and coping with minority stress can affect key psychosocial outcomes, such as coping self-efficacy and symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 13-19 years of age (inclusive)
2. Self-identify as a sexual or gender minority
3. Are English literate
4. Reside within the United States
5. Have access to a device that has internet access, a web browser, and SMS capabilities, such as a smartphone, computer, or tablet
6. Willingness to participate in study activities

Exclusion Criteria:

1. Not between 13-19 years of age (inclusive)
2. Does not self-identify as a sexual or gender minority
3. Is not English literate
4. Does not reside within the United States
5. Does not have access to a device that has internet access, a web browser, and SMS capabilities, such as a smartphone, computer, or tablet
6. Unwilling to participate in study activities

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Bauermeister, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Study variables will be available; however, the investigators will protect the rights and privacy of human subjects by redacting all identifiers from the dataset.
Supporting Information: Study Protocol, SAP
Time Frame: The investigators will assure the timely release and sharing of data two years after the publication of the main trial findings from the final dataset.
Access Criteria: The de-identified data from this project will be available through individual requests directed to the Principal Investigator.

REFERENCES:
- [Derived] Bauermeister J, Choi SK, Bruehlman-Senecal E, Golinkoff J, Taboada A, Lavra J, Ramazzini L, Dillon F, Haritatos J. An Identity-Affirming Web Application to Help Sexual and Gender Minority Youth Cope With Minority Stress: Pilot Randomized Controlled Trial. J Med Internet Res. 2022 Aug 1;24(8):e39094. doi: 10.2196/39094. PMID 35916700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Online Resource Website | Immi
Started | 135 | 135
Completed | 122 | 122
Not Completed | 13 | 13
Not completed — Lost to Follow-up | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Resource Website | Immi | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 120 | 123 | 243
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.42 (1.51) | 16.56 (1.46) | 16.49 (1.49)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Multiple gender identities | 56 | 57 | 113
  Single gender identity | 79 | 78 | 157
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 106 | 209
  Male | 32 | 29 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 31 | 73
  Not Hispanic or Latino | 93 | 104 | 197
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 23 | 26 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 23 | 42
  White | 28 | 32 | 60
  More than one race | 64 | 54 | 118
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 135 | 135 | 270

OUTCOME MEASURES:

1. Primary Outcome: Coping Self-efficacy
Description: The Stress Appraisals Measure for Adolescents includes three subscales (Challenge subscale; Threat subscale; Resources subscale). Each of these subscales is answered on a 5-point scale (1=strongly disagree to 5=strongly agree). A mean score was computed for each subscale, with higher values indicating greater endorsement of each respective stress appraisal.
Time Frame: 4-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Resource Website | Immi
Number analyzed (Participants) | 122 | 122
score on a scale
  Challenge | 3.32 (.93) | 3.64 (.85)
  Threat | 3.92 (.69) | 3.85 (.77)
  Resource | 3.67 (.90) | 3.83 (.92)

2. Secondary Outcome: Identity Affirmation
Description: The Lesbian, Gay and Bisexual Positive Identity Measure-Authenticity Subscale has a scoring range from 1 to 7 (1=strongly disagree to 7=strongly agree). A mean score was computed, whereby greater values indicate greater feelings of authenticity.
Time Frame: 4-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Resource Website | Immi
Number analyzed (Participants) | 122 | 122
units on a scale | 5.08 (1.30) | 5.10 (1.33)

3. Secondary Outcome: Internalization of Minority Stress
Description: The Coping with Discrimination Scale- Internalization Subscale has a scoring range from 1 to 6 (1=never to 6=always). We computed a mean score, where higher scores indicate greater internalization of blame for minority stress
Time Frame: 4-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Resource Website | Immi
Number analyzed (Participants) | 122 | 122
score on a scale | 2.94 (1.23) | 3.19 (1.27)

4. Secondary Outcome: Sense of Belonging to the Queer Community
Description: The Thwarted Belongingness subscale of the Interpersonal Needs Questionnaire is a 5-item scale that is answered on a 7-point scale (1=not at all true" to 7=very true for me). We computed a sum score ranging from 5 to 35, where higher scores indicate a lack of sense of belonging
Time Frame: 4-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Resource Website | Immi
Number analyzed (Participants) | 122 | 122
units on a scale | 18.21 (6.24) | 17.15 (6.99)

5. Secondary Outcome: Anxiety Symptoms
Description: The General Anxiety Disorder-7 scale has a range from 0 to 21. Scores were computed by summing the items. Higher scores indicate greater anxiety symptomatology.
Time Frame: 4-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Resource Website | Immi
Number analyzed (Participants) | 122 | 122
score on a scale | 10.30 (5.78) | 9.92 (5.56)

6. Secondary Outcome: Depression Symptoms
Description: The Patient Health Questionnaire-8 inventory has a range from 0 to 24. A summed score was computed, where higher scores indicate greater depression symptomatology.
Time Frame: 4-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online Resource Website | Immi
Number analyzed (Participants) | 122 | 122
score on a scale | 11.40 (5.75) | 11.61 (5.95)

7. Secondary Outcome: Cognitive and Behavioral Coping Skills
Description: The Brief COPE inventory is comprised of 11 subscales: Self-distraction; Active coping; Emotional support; Instrumental support; Venting; Positive reframing; Planning; Acceptance; Self-blame; Substance use; and, Behavioral disengagement. Participants answered each subscale using a 4-point scale (1="I haven't been doing this at all" to 4="I've been doing this a lot"). A mean score was computed for each subscale, with higher values indicating greater use of that coping skill.
Time Frame: 4-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Online Resource Website | Immi
Number analyzed (Participants) | 122 | 122
units on a scale
  Self-distraction | 3.23 (.65) | 3.23 (.65)
  Active coping | 2.47 (.72) | 2.65 (.84)
  Emotional support | 2.43 (.94) | 2.59 (.94)
  Instrumental support | 2.30 (.87) | 2.64 (.90)
  Venting | 2.42 (.82) | 2.48 (.86)
  Positive reframing | 2.25 (.78) | 2.45 (.86)
  Planning | 2.56 (.86) | 2.79 (.83)
  Acceptance | 2.73 (.77) | 2.87 (.77)
  Self-blame | 2.76 (.88) | 2.91 (.87)
  Substance use | 1.38 (.78) | 1.33 (.74)
  Behavioral disengagement | 1.99 (.82) | 2.01 (.80)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Online Resource Website | Immi
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/135
Other Adverse Events (participants affected / at risk) | 0/135 | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT05061966/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT05061966/ICF_001.pdf